CLINICAL TRIAL: NCT05453513
Title: The Neural Underpinnings of Depression and Cannabis Use in Young People Living With HIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Vilma Gabbay, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20230798; R01DA054885 (NIH)
Record Dates: First submitted 2022-07-01; First posted 2022-07-12 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-05

CONDITIONS: Depression; Cannabis Use Disorder; HIV
MeSH Terms: conditions — Depression

STUDY DESIGN:
Masking Description: No masking, all participants will undergo the same procedures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neural Underpinnings of Depression Group (Experimental): All participants will undergo neuroimaging and behavioral tests. during the course of the study (12 months).
  Interventions: Behavioral: MRI Study

INTERVENTIONS:
Behavioral: MRI Study — fMRI Tasks

SUMMARY:
To elucidate mechanisms of substance use disorders (SUD) and comorbid mental illnesses in people living with HIV (PLWH), the study team seeks to investigate reward and pain circuitry in cannabis use and depression comorbidity, two highly prevalent conditions in PLWH. The study team proposes a tightly integrative study to test the overall hypothesis that cannabis use and depression in young PLWH have an additive effect, inducing both reward deficits and pain hypersensitivity, and that this pattern will predict worse outcomes at 1 year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositivity confirmed with lab report, medical records, or HIV testing.
* Between the ages of 18-39 years
* Fluency in English or Spanish
* Ability to provide informed consent and perform study procedures, including estimated full-scale intelligence quotient (IQ) >75 to ensure that participants are able to understand the study.
* Cannabis users: To capture a wide range of cannabis use frequency, meeting Diagnostic and Statistical Manual 5 (DSM-5) criteria for Cannabis use Disorder (CUD) will not be required. However, in order to ensure sufficient exposure, cannabis use will be significant (self-reported use on ≥20 of the prior 30 days and positive THC urine toxicology).
* Depressed: In order to capture a wide range of depression illness severity, we will allow participants with subthreshold depression, defined as a raw severity score of ≥12 on the Montgomery Asberg Depression Rating Scale (MADRS).

Exclusion Criteria:

* Perinatally acquired HIV infection, as early neurodevelopmental alterations and HIV legacy effects may exist in this group
* Pregnancy or lactation
* Current Substance Use Disorder other than cannabis or nicotine
* Certified for or self-reported medical cannabis use, or intent to become certified
* Current cocaine use by self-report or urine toxicology
* central nervous system (CNS) disease or injury, or neuro-degenerative disease
* Unique pain syndromes (e.g. multiple sclerosis, rheumatoid arthritis);
* Severe medical illness such as end-stage renal disease, heart failure, cirrhosis, or cancer
* MRI contraindication such as claustrophobia, metallic ink tattoos, or pacemaker.

Depressed cannabis non-users:

* At baseline, all participants will be psychotropic-medication-free for ≥1 month prior to study enrollment (or ≥3 months for medications with longer half-lives). Benzodiazepines and sleeping aids taken on an as-needed basis will be allowed, however we will require a 4-day abstinence period before the scan.
* Exclusionary are participants with a DSM-5 diagnoses of bipolar disorder, psychotic disorders, autism spectrum disorders, and all non-cannabis substance-related disorders will be exclusionary. disorder (PTSD) are not uncommon among depressed individuals and will be
* Anxiety disorders, obsessive-compulsive disorder (OCD), and post-traumatic stress are allowed as long as depressive symptoms are primary.

atypical of depression. • Suicidal ideations (SI) without a specific plan (defined as passive SI) are common in depression and will be allowed. However, if SI constitutes an imminent risk to self or others (defined as active SI), the participant will be withdrawn from the study and emergency procedures will be initiated immediately, including ER admission.

Depressed cannabis users:

• Exclusion criteria will be the same as depressed cannabis non-users except for cannabis use.

Non-depressed cannabis users:

• Will have no major psychiatric conditions other than cannabis use/disorder.

Non-depressed cannabis non-users:

• Exclusion criteria will be the same as for non-depressed cannabis users; in addition participants will not report cannabis use in the prior 90 days and have a urine toxicology test negative for cannabis.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Addiction Severity Index (ASI) | Up to 1 year
  The number of days using illicit opioids in the past 30 days per self-report as collected through the Addiction Severity Index.
Montgomery Asberg Depression Rating Scale (MADRS) Scale | Up to 12 months
  Measures the severity of depressive episodes in patients with mood disorders Scale 0-60 higher more severe
Temporal Experience of Pleasure Scale (TEPS) | Up to 12 months
  Self-report measure allowing the assessment of anticipatory and consummatory pleasure 25 to 120 higher more pleasure
Neural Circuitry measured by MRI | Baseline
  Measured using Magnetic Resonance Imaging. Summary beta values representing the level of brain activity will be calculated.

SECONDARY OUTCOMES:
Daily Sessions Frequency Age Quantity of Cannabis Use Inventory (DFAQ- CU) | Up to 12 months
  Measures cannabis consumption Score range 0 to 185. The higher the score, the greater the usage of cannabis.
Timeline Followback (TLFB) | Up to 12 months
  Tool to obtain a variety of estimates of marijuana, cigarette, and other drug use. scores range from days of use (0-30)
tetrahydrocannabinol (THC) Metabolite, Serum | Up to 12 months
  Suggests use of, or exposure to, a product containing THC. pmol/mL
Fagerström Test for Nicotine Dependence full-term normal delivery (FTND) | Up to 12 months
  The FTND is a validated, 6-item self-report instrument that evaluates the intensity of physical addiction to nicotine. Three items are rated yes/no (0/1), and the other three items are rated on a scale from 0-3. Items are summed to yield a total score of 0-10, with higher scores reflecting greater nicotine dependence.
Beck Depression Inventory-II (BDI-II) | Up to 12 months
  Designed to assess the presence and severity of depressive symptoms Score 0-63 higher the score greater the depression
Snaith-Hamilton Pleasure Scale (SHAPS) | Up to 12 months
  Measures anhedonia, the inability to experience pleasure Score 0-42 greater the score greater the pleasure.
Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) | Up to 12 months
  Alcohol consumption will be measured using total score on the 3-item Alcohol Use Disorders Identification Test-Consumption (AUDIT-C) which includes typical quantity and frequency, and frequency of binge drinking (# of drinks modified by age based on the NIAAA Youth Guide). Higher score indicates worse outcomes.
Cannabis Use Problem Identification Test (CUPIT) | Up to 12 months
  6-item self-reported questionnaire assessing cannabis use and dependence; Range 3-82, higher values indicating a more severe cannabis use disorder.
Pittsburgh sleep quality index | up to 12 months
  Assesses sleep quality and disturbances over a month period Scores 0-24 higher the score greater sleep dysfunction
Brief Pain Inventory (BPI) | up to 12 months
  Assesses the severity of pain and its impact on functioning. Pain questionnaire (0-10; higher score=worse)
Pain Anxiety Symptom Scale (PASS-20) | up to 12 months
  Measures fear and anxiety responses specific to pain Range 0-100 higher the more anxiety symptoms
HIV RNA test | Baseline
  HIV RNA test detects HIV and not antibodies 20 to 10,000,000 copies/mL higher the amount the more infectious
cluster of differentiation 4 (CD4+) / cluster of differentiation 8 (CD8+) | Up to 12 months
  Monitors the immune system Flow cytometry will be used to detect serum CD4, CD8
HIV Visual Analogue Scale (HIV-VAS) | 12 month
  The VAS asks individuals to mark a line at the point along a continuum showing how much of each drug they have taken in the last 4 weeks 0-30 higher score worse pain

CONTACTS AND LOCATIONS:
Overall Officials: Vilma Gabbay, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No